CLINICAL TRIAL: NCT00512954
Title: A Prospective One Year Study of the Causes, Characteristics, Mechanisms and Kinetics of Exacerbations in Subjects With Asthma
Brief Title: Causes, Characteristics and Mechanisms of Infective Exacerbations in Subjects With Asthma and Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: GlaxoSmithKline (Industry); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Parameswaran Nair, McMaster University, Firestone Institute for Respiratory Health
Other Study IDs: 06-2671
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-07

CONDITIONS: Asthma; COPD
Keywords: airway inflammation; susceptibility to infections; inflammatory response in blood and urine; infective exacerbations; asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diseases of the airways (bronchi) of the lungs include asthma and chronic obstructive pulmonary disease (COPD), which are leading causes of reduced quality of life, loss of work, hospital admissions and deaths and result in a major economic burden to the patient and society. Worsening (exacerbation) of these conditions is common and is frequently due to viral or bacterial infection, which causes inflammation in the bronchi, i.e. bronchitis. Ways to objectively measure the inflammation are needed to improve diagnosis, cause and severity and to guide treatment. The investigators also need to understand changes in the body's defense (immune) mechanisms that make some patients have more frequent infective bronchitis.

At present, sputum cell counts are able to identify different types of bronchitis, their severity and may be able to differentiate viral from bacterial infection. Other measurements in sputum, exhaled breath, blood and urine are also available to measure this inflammation. Measurement of immune cells in the blood gives us an idea about the working capacity of the immune system of the body.

The investigators plan to study patients with asthma or COPD at the time of worsening of their condition to identify,

1. To what extent viral or bacterial bronchitis can be diagnosed from tests of inflammation?
2. How clearing of infection relates to clearing of inflammation?
3. What are the changes in the body's defense mechanisms that make a patient more prone to frequent infective bronchitis?
4. How do the measurements in sputum, exhaled breath, blood and urine relate to viral and bacterial bronchitis?
5. What are the differences in the measurements in sputum, exhaled breath, blood and urine in asthma and COPD?

DETAILED DESCRIPTION:
Exacerbations of asthma and COPD are a major cause of morbidity, mortality and economic burden to the patient and society. Exacerbations are usually associated with worsening of airway inflammation which, as identified by quantitative sputum cell counts, can be neutrophilic, eosinophilic, combined eosinophilic and neutrophilic or neither, a result of different causes. The commonest cause of exacerbations is infection. Neutrophilic exacerbations are common and are usually associated with bacterial and non-bacterial infections but eosinophilic exacerbations might also predict viral infections. However the investigators are still unsure whether aspects of neutrophilic inflammation can differentiate viral from bacterial infections. Also the exact relationship between etiology, mechanisms of susceptibility to infection, inflammation and airway responsiveness during an exacerbation is poorly understood. As a result, the physician assumes that clinical improvement from an exacerbation corresponds to resolution of infection and underlying inflammation of airways at the same time. However, inflammation of the airways may persist beyond the resolution of infection, which may contribute to the morbidity and mortality of the disease.

The primary objective of this study is to better understand the correlation between the different types of inflammation and infection of the airways during exacerbations. Secondary objectives are to understand the susceptibility to infections and methods to assess the inflammatory response and airway responsiveness during infections. To attain these objectives we will compare the total cells, percentage of neutrophils, percentage of eosinophils in sputum and nasal secretions, sputum fibrinogen, sputum total lactate dehydrogenase, microbial load in sputum and nasal secretions, exhaled nitric oxide, p H of exhaled breath condensate, serum procalcitonin, intensity of urinary 3-bromotyrosine, 3-chlorotyrosine, 3, 5- dibromotyrosine and dityrosine, symptom score, FEV1 and Mannitol PD15 at different time points during an exacerbation, compare the activity of toll like receptors (2,4,7,9) and natural killer T cells during the stable phase of disease with the number of infective exacerbations during the course of one year and test the feasibility of mannitol challenge testing as a method to induce sputum and measure airway hyperresponsiveness. Our approach will be to identify 100 patients with variable (asthma) or chronic airflow limitation (COPD), reporting within 2 to 5 days of the onset of an exacerbation during the course of one year. The clinical, physiological, inflammatory, microbiological and immunological parameters will be assessed on the day of presentation (day 0), day 7, 14 and at 6 to 8 weeks. The information collected at 6 to 8 weeks will serve as baseline data, if the patient is clinically stable at this point in time. If the patient has a next exacerbation during the course of the trial, then the same procedure will be followed.

This work will enhance the knowledge of issues needed to improve diagnosis of exacerbations of airways disease, their causes, the mechanisms involved and the most appropriate treatment. The results may lead to future randomized controlled trials, in which treatment of exacerbations will be based on the most appropriate measurements that will eventually lead to better management of airway diseases, reduce the overall cost of therapy and improve the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (medically or surgically postmenopausal or practicing an accepted form of barrier or hormonal contraception) subjects between 18 - 80 years.
2. Any severity of exacerbation of obstructive airway disease attending the outpatient clinic.
3. History of at least two exacerbations in the past 12 months prior to recruitment that required a course of prednisone or antibiotic or long acting bronchodilator or inhaled corticosteroid, in addition to the daily maintenance therapy.
4. Signed written informed consent to participate in the protocol and ability to return to the outpatient clinic for repeated clinic visits.

Exclusion Criteria:

1. If the exacerbation is severe enough to warrant hospitalization.
2. Active malignancy.
3. Significant gastrointestinal, hematological, cardiovascular or cerebrovascular disorder that would affect compliance with follow up visits.
4. Recent (within the past 2 months) or planned (within the study period) lung surgery.
5. Psychosis, alcoholism, active substance abuse or any personality disorder that would make compliance with the follow up visits problematic.
6. Pregnant or nursing females, as this could affect the compliance during the trial.
7. Any other medical or social condition, which in the opinion of the investigator could confound the interpretation of the data derived from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatics with 1 or more exacerbation in last calendar year.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran K Nair, MD, PhD, Principal Investigator — Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario; Frederick E Hargreave, MD, Principal Investigator — Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Jayaram L, Pizzichini MM, Cook RJ, Boulet LP, Lemiere C, Pizzichini E, Cartier A, Hussack P, Goldsmith CH, Laviolette M, Parameswaran K, Hargreave FE. Determining asthma treatment by monitoring sputum cell counts: effect on exacerbations. Eur Respir J. 2006 Mar;27(3):483-94. doi: 10.1183/09031936.06.00137704. PMID 16507847
- [Background] Johnston SL. Overview of virus-induced airway disease. Proc Am Thorac Soc. 2005;2(2):150-6. doi: 10.1513/pats.200502-018AW. PMID 16113484
- [Background] Papi A, Bellettato CM, Braccioni F, Romagnoli M, Casolari P, Caramori G, Fabbri LM, Johnston SL. Infections and airway inflammation in chronic obstructive pulmonary disease severe exacerbations. Am J Respir Crit Care Med. 2006 May 15;173(10):1114-21. doi: 10.1164/rccm.200506-859OC. Epub 2006 Feb 16. PMID 16484677
- [Background] Chaudhuri N, Dower SK, Whyte MK, Sabroe I. Toll-like receptors and chronic lung disease. Clin Sci (Lond). 2005 Aug;109(2):125-33. doi: 10.1042/CS20050044. PMID 16033327
- [Background] Akbari O, Faul JL, Hoyte EG, Berry GJ, Wahlstrom J, Kronenberg M, DeKruyff RH, Umetsu DT. CD4+ invariant T-cell-receptor+ natural killer T cells in bronchial asthma. N Engl J Med. 2006 Mar 16;354(11):1117-29. doi: 10.1056/NEJMoa053614. PMID 16540612
- [Background] Silkoff PE, Carlson M, Bourke T, Katial R, Ogren E, Szefler SJ. The Aerocrine exhaled nitric oxide monitoring system NIOX is cleared by the US Food and Drug Administration for monitoring therapy in asthma. J Allergy Clin Immunol. 2004 Nov;114(5):1241-56. doi: 10.1016/j.jaci.2004.08.042. PMID 15536442
- [Background] Simon L, Gauvin F, Amre DK, Saint-Louis P, Lacroix J. Serum procalcitonin and C-reactive protein levels as markers of bacterial infection: a systematic review and meta-analysis. Clin Infect Dis. 2004 Jul 15;39(2):206-17. doi: 10.1086/421997. Epub 2004 Jul 2. PMID 15307030
- [Background] Leuppi JD, Salome CM, Jenkins CR, Anderson SD, Xuan W, Marks GB, Koskela H, Brannan JD, Freed R, Andersson M, Chan HK, Woolcock AJ. Predictive markers of asthma exacerbation during stepwise dose reduction of inhaled corticosteroids. Am J Respir Crit Care Med. 2001 Feb;163(2):406-12. doi: 10.1164/ajrccm.163.2.9912091. PMID 11179114
- [Background] Kharitonov SA, Barnes PJ. Exhaled biomarkers. Chest. 2006 Nov;130(5):1541-6. doi: 10.1378/chest.130.5.1541. PMID 17099035